CLINICAL TRIAL: NCT03166800
Title: MitoQ for Fatigue in Multiple Sclerosis: a Placebo Controlled Trial
Brief Title: MitoQ for Fatigue in Multiple Sclerosis
Acronym: MS
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of adequate funding
Sponsor: Oregon Health and Science University (Other)
Collaborators: MitoQ Limited (Unknown); National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Vijayshree Yadav, MD, MCR, FANA, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00015779
Record Dates: First submitted 2017-05-23; First posted 2017-05-25 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Multiple Sclerosis; Fatigue
Keywords: mitoquinone; Fatigue; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis; Fatigue | interventions — mitoquinone; mitoquinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): 20 subjects will receive placebo.
  Interventions: Drug: Placebo
- 20mg oral MitoQ (Active Comparator): MitoQ is a potent antioxidant supplement with potentially significant immunomodulatory and anti-inflammatory properties. 20mg of MitoQ will be administered to 20 subjects in this trial.
  Interventions: Drug: Mitoquinone
- 40mg oral MitoQ (Active Comparator): MitoQ is a potent antioxidant supplement with potentially significant immunomodulatory and anti-inflammatory properties. 40mg of MitoQ will be administered to 20 subjects in this trial.
  Interventions: Drug: Mitoquinone

INTERVENTIONS:
Drug: Mitoquinone — This arm of the intervention the study subject will be administered 40mg of the study drug MitoQ orally in capsule form every morning for 12 weeks.
  Other Names: mitoquinol
  Arms: 40mg oral MitoQ
Drug: Mitoquinone — This arm of the intervention the study subject will be administered 20mg of the study drug MitoQ orally in capsule form every morning for 12 weeks.
  Other Names: mitoquinol
  Arms: 20mg oral MitoQ
Drug: Placebo — This arm of the intervention the study subject will be administered placebo capsules to orally take every morning for 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether MS patients who receive Oral mitoquinone (MitoQ) have less fatigue than those receiving a placebo. A comparison between patient's fatigue scored at baseline and fatigue scored 12 weeks after study drug initiation will assess if MitoQ has a significant change in fatigue.

DETAILED DESCRIPTION:
MitoQ is a potent antioxidant with potentially significant immunomodulatory and anti-inflammatory properties. While the cause of MS related fatigue is uncertain, the investigators believe that mitochondria dysfunction and resultant neuronal energy depletion may be an important contributor to fatigue in MS.

This clinical trial will evaluate the potential beneficial effects of MitoQ on MS fatigue. It will also explore the effects of MitoQ on cognitive function, quality of life and mood. If enrolled in the study, patients will take two capsules of the study drug or placebo at the same time every day for twelve weeks. There will be 4 study visits where the participant will undergo medical and nervous system examinations, questionnaires, and blood draws. Because it is a placebo-controlled trial, participants will have a 33% chance of receiving either placebo (inactive), 20mg of MitoQ, or 40mg of MitoQ. This will be a blinded randomized study, meaning neither the participant nor the investigator will know who received the placebo or study drug.

ELIGIBILITY:
Inclusion Criteria:

* MS (any clinical subtype) as diagnosed by the 2010 McDonald criteria40;
* Expanded Disability Status Scale (EDSS) score of 2 to 8,
* Complaint of fatigue that has been persistent for at least two months;
* Modified Fatigue Impact Scale (MFIS) score of 38 or greater

Exclusion Criteria:

* Treatment with systemic glucocorticoids in the prior six weeks;
* Beck Depression Inventory (BDI) >31 (severe depression);
* Significant MS exacerbation in prior 30 days;
* Previous use of MitoQ or CoQ-10 within 30 days of screening appointment;
* Use of non-research-pharmacy-administered MitoQ or CoQ-10 during the duration of the study;
* Other significant health problem (e.g. active coronary heart disease, liver disease, pulmonary disease, diabetes mellitus) that might increase risk of patient experiencing adverse events),
* Pregnancy or intending to become pregnant or breastfeeding;
* Unable to complete the self-report forms;
* Unable to give informed consent;
* Prisoners will be excluded.
* Any condition which would make the patient, in the opinion of the investigator, unsuitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Fatigue measured by Modified Fatigue Impact Scale (MFIS) Score at 12 weeks post study drug initiation | Baseline to 12 weeks post drug initiation.
  This primary outcome measure will be the difference from baseline in fatigue scores as measured by Modified Fatigue Impact Scale (MFIS) Score at 12 weeks post study drug initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Vijayshree Yadav, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided